CLINICAL TRIAL: NCT05230797
Title: Clinical and Radiographic Evaluation of Zinc Oxide-Propolis Versus Zinc Oxide- Eugenol as Obturating Material in Primary Teeth Pulpectomy: A Randomized Clinical Trial
Brief Title: Zincoxide-propolis vs Zincoxide-eugenol Pulpectomy
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nora Ahmed Kadry, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZOP pulpectomy
Record Dates: First submitted 2021-11-30; First posted 2022-02-09 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Pulp Necroses
MeSH Terms: conditions — Dental Pulp Necrosis | interventions — Zinc Oxide-Eugenol Cement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- zinc-oxide propolis (Experimental): Propolis is a natural resinous mixture produced by honeybees from substances collected from parts of plants, buds, and exudates. The essential principle compounds responsible for biological activities are polyphenols, aromatic acids, and diterpenic acids. Numerous biological properties of propolis have been reported including cytotoxic, antiherpes, free radical scavenging, antimicrobial, and anti-HIV activities The antibacterial effect of propolis is bactericidal by inhibiting their mobility. Propolis kills the fungi and also inhibits the growth of the viruses.
  Interventions: Drug: Zinc oxide Propolis
- zinc-oxide eugenol (Active Comparator): Zinc oxide-eugenol cement (ZOE) has been used as a root canal filling material for primary teeth and has long been the material of choice of pediatric dentists worldwide, although it fails to meet the ideal requirements of root canal filling material for primary teeth due to limited antimicrobial action, and a slower rate of resorption than the roots of the primary teeth. Studies report that the success rate of ZOE ranges from 65% to 86% so it's materials of choice if primary teeth are not nearing exfoliation.
  Interventions: Drug: Zinc Oxide-Eugenol Cement

INTERVENTIONS:
Drug: Zinc oxide Propolis — antibacterial and anti-inflammatory
  Other Names: Also called Bee wax
  Arms: zinc-oxide propolis
Drug: Zinc Oxide-Eugenol Cement — Antimicrobial and antiseptic
  Other Names: ZOE
  Arms: zinc-oxide eugenol

SUMMARY:
The clinical trial aims to evaluate the clinical and radiographic success of Zinc oxide- propolis versus Zinc oxide -Eugenol as obturating material in pulpectomy of non-vital primary teeth.

DETAILED DESCRIPTION:
Pulpectomy is considered the most convenient way to treat the non-vital primary teeth as it preserves the affected tooth to maintain the length and integrity of the dental arch until exfoliation4. Zinc oxide-eugenol cement (ZOE) has been used as a root canal filling material for primary teeth and has long been the material of choice of pediatric dentists worldwide, although it fails to meet the ideal requirements of root canal filling material for primary teeth due to limited antimicrobial action, and a slower rate of resorption than the roots of the primary teeth. Concerns about these drawbacks of ZOE directed to search for alternative obturating materials for primary teeth.

Propolis, a natural resinous substance, is collected by honey bees with potent antimicrobial and anti-inflammatory properties. The main chemical constituents present in propolis are flavonoids, phenolics, and other aromatic compounds. Considering these beneficial effects of propolis, a zinc oxide-propolis mixture is suggested to increase the survival rate and improve the treatment prognosis of non-vital primary teeth.

ELIGIBILITY:
Inclusion Criteria:

* Children 4-6 years
* Non-vital primary molars
* Teeth with radiographic evidence of minimum bone loss.

Exclusion Criteria:

* Primary molars with less than two-thirds of the remaining root length
* Molars demonstrating extensive external or internal resorption,
* Teeth exhibiting greater than Grade I mobility
* Non-restorable with stainless steel
* Children whose parents or caregivers did not give consent for the study

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-08 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Absence of Pain | 9 months
  •Measuring Method : Verbal Question to Patient /Parents
  •Measuring Unite: Binary